CLINICAL TRIAL: NCT03786055
Title: Impact of Somatic Yoga and Meditation on Fall Risk, Function, and Quality of Life for Chemotherapy-Induced Peripheral Neuropathy Syndrome in Cancer Survivors
Brief Title: Somatic Yoga and Meditation for Cancer Survivors With Pain From Neuropathy
Acronym: Y4CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockton University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.019
Record Dates: First submitted 2018-11-21; First posted 2018-12-24 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Cancer Survivor; Pain; Chemotherapy Induced Peripheral Neuropathy; Function; Fall Risk; Balance; Quality of Life
Keywords: cancer survivor; pain; chemotherapy induced peripheral neuropathy; fall risk; quality of life; somatic yoga; meditation
MeSH Terms: conditions — Pain | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Criteria for enrollment included cancer survivors age 18 or older; any type or stage of cancer, currently completed all treatment with no current evidence of disease; at least mild peripheral neuropathy symptoms (either sensory or motor) as rated on the Patient Neurotoxicity Questionnaire (PNQ), attributable to chemotherapy intervention as a component of cancer treatment. Exclusion criteria included active cancer disease or current cancer treatment; co-morbidities such a diabetes or prior history of peripheral neuropathy from any cause. All participants will be screened with the physical activity readiness questionnaire (PAR-Q) to determine the safety or possible risk of exercising based on health history, current symptoms and risk factors. Somatic yoga and meditation (SYM) will be provided during 16 sessions/8 weeks for 1.5 hours and participants will complete home-based SYM and journal entries.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Somatic Yoga and Meditation (SYM) (Experimental): Participants will engage in 16 sessions of somatic yoga and meditation with appropriate props as needed over 8 weeks and continue with a home practice. Application of SYM throughout activities of daily living is reinforced. All sessions are facilitated by trained yoga therapists.
  Interventions: Behavioral: Somatic Yoga and Meditation (SYM)

INTERVENTIONS:
Behavioral: Somatic Yoga and Meditation (SYM) — A Hanna somatics and somatic yoga and meditation (SYM) protocol was designed to address sensory-motor amnesia and reduce trauma which creates reflex patterns that lead to chronic muscular contractions. The movements use voluntary muscular contraction and slow controlled eccentric contraction, with the constant focus on sensation to increase the resting length of muscles. Movements are performed slowly and gently with the least possible effort and are never forced. The protocol is endorsed by the US Army Surgeon General as treatment for chronic pain. The meditations are trauma informed and evidence based supporting pain modulation, healing and well-being.
  Other Names: Yoga4CIPN (Y4CIPN)

SUMMARY:
Chemotherapy-induced peripheral neuropathy syndrome (CIPN) causes significant pain in hands and feet and is an adverse effect of treatment. Few non-pharmacological interventions have been tested and individuals experience CIPN symptoms years after treatment. This is the first study to explore a somatic yoga and meditation (SYM) intervention on functional outcomes and quality of life in cancer survivors.

DETAILED DESCRIPTION:
Pain is a common symptom associated with cancer; 75-90% of cancer patients experience pain during their illness and up to 50% of that pain is undertreated. Unrelieved pain leads to increased levels of the stress hormone cortisol. Chemotherapy-induced peripheral neuropathy syndrome (CIPN) causes significant pain in hands and feet and is a common, adverse effect of several chemotherapeutic agents. It can lead to abrupt discontinuation of treatment, and severely affects the quality of life.

CIPN is a particularly important adverse effect because it may compromise the ability to tolerate chemotherapy and become a serious, long-lasting, and even permanent debility. CIPN symptoms may persist many years after treatment; together with worse function, greater disability, and more falls which is complicated by the aging process. Clinically, CIPN presents as deficits in sensory, motor, and function which develop in a glove and stocking distribution.

While chemotherapy improves the likelihood of disease-free survival, the result of CIPN may cause decreased walking speed and balance observed after the first chemotherapy cycle and progresses with cumulative exposure. These functional deficits are mirrored with increased symptom severity. CIPN is associated with potential fall risk with aging cancer survivors and increased functional disability.

Few interventions have been tested for impact from CIPN. Yoga is a popular movement therapy, often used by cancer survivors for symptom management. Several studies demonstrate the promising effects of yoga on sleep, fatigue and quality of life (QOL) in cancer survivors. However, no study has rigorously investigated its effects on CIPN and quality of life.

This study will explore the preliminary therapeutic effects of an 8-week somatic based yoga and meditation (SYM) program and 15-25 cancer survivors with CIPN will be enrolled into a small pilot study. This will include 16 sessions of yoga designed specifically to minimize injury, promote flexibility/ balance and to allow you to maximize their specific functional goals. All types of cancer diagnoses resulting in CIPN will be enrolled in a single arm feasibility trial. SYM will be provided twice a week for 8 weeks for 1.5 hours. You will complete surveys at the beginning and end of 8 weeks and receive a home-based SYM and write journal entries to determine your perspectives of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors 18 years or older
* Any type or stage of cancer
* Completed chemotherapy treatment
* Mild Peripheral Neuropathy Symptoms

Exclusion Criteria:

* Active cancer disease
* Currently receiving cancer treatment
* Diabetes
* Prior history of peripheral neuropathy from other disease
* Risk factors for exercise (measured by Patient Activity Readiness Questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Sit and Reach (SR) | Change from baseline flexibility at 8 weeks
  The Sit and Reach Test (SR) is the most-widely used measure of hamstring and low back flexibility, examining the maximal reach an individual can make in a long-sitting position. The SR has established norms by the American College of Sports Medicine, with a score of 16 and 15 for adults 46-55 years old and 56-65 years old respectively in the 50th percentile. Individuals are asked to maintain a long-sit position on the floor while safely reaching forward as far as possible with their shoes removed, feet flat against the table, and legs straight. Three trials are averaged and higher scores indicate greater flexibility.
Forward Reach (FR) | Change from baseline balance at 8 weeks
  The Functional Reach test (FR) test examines the balance of individuals with respect to the patient's limit of stability. Each participant is instructed to flex the test arm forward to 90˚ and to reach forward as far as possible before taking a step. The reach is determined by the total excursion of the third metacarpal from the starting point to the point just before balance is lost. An average of 3 measurements is used as the final score. FR has demonstrated strong reliability and validity for measuring postural control in reaching forward during standing. The FR test has shown criterion validity, predictive validity, test-retest reliability, and inter-rater reliability for younger and older adults. It has also been shown to possess predictive validity for falls.
Timed Up and Go (TUG) | Change from baseline walking speed at 8 weeks
  The Timed Up and Go (TUG) is a standardized test that measures physical function in sitting to standing, walking and returning to the seated position. Participants are instructed to stand up from a chair, walk three meters as quickly and safely as possible, turn around, walk back and sit down. The test is timed and longer time indicates worse performance. Nine seconds is the cutoff for high risk of falls.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | Change from baseline pain at 8 weeks
  The BPI is a patient reported outcome measure that assesses severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. It responds to both behavioral and pharmacological pain interventions and takes 5 minutes to complete. Scoring algorithm: "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference. Reliability: Cronbach alpha reliability ranges from 0.77 to 0.91
Patient Neurotoxicity Scale (PNQ) | Change from baseline sensation and strength at 8 weeks
  Patient perception of sensation and weakness attributed to CIPN.The PNQ is two self-reflective questions and quantifies the symptoms (sensation) and perceived weakness from CIPN 1) Do you have numbness, pain, or tingling in your hands or feet? 2) Do you have weakness in your arms or legs? These two items are rated 1-5 on the following scale: 1 = No, 2 = Mild, 3 = Moderate, 4 = Moderate-to-Severe, and 5 = Severe. The PNQ total score ranges from 2 to 10, with a high total score indicating severe CIPN symptoms. A PNQ total score of 2 is defined as grade A; 3-4, as grade B; 5-6, as grade C; 7-8, as grade D; and 9-10, as grade E
Perceived Stress Scale (PSS) | Change from baseline stress at 8 weeks
  Each item is rated on a 5-point scale ranging from never (0) to almost always (4). Positively worded items are reverse scored, and the ratings are summed, with higher scores indicating more perceived stress. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. ► Scores ranging from 0-13=low stress. ► Scores ranging from 14-26 = moderate stress. ► Scores ranging from 27-40 = high perceived stress.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline sleep at 8 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (Fact/GOG-Ntx) | Change from baseline quality of life at 8 weeks
  The FACT/GOG-Ntx contains 11 items scored from 0-4, and scores are summed for a range of 11-44. Questions on the Ntx subscale pertain to the feeling of weakness all over, numbness or tingling in the hands or feet, and difficulty buttoning their buttons. Reliability was measured using Cronbach alpha of greater than 0.7 and higher scores indicate greater severity of symptoms.
Falls Efficacy Scale (FES) | Change from baseline fear of falling at 8 weeks
  The FES is a 10 item scale where each item is rated on a scale of 1-10. A score of 10 signifies no confidence in these activities; a score of 1 indicates confidence. Out of a total score of 100, a score of 70 or above indicates the individual has a fear of falling.

OTHER OUTCOMES:
Vibration Sense - Biothesiometer | Change from baseline sensation at 8 weeks
  A calibrated biothesiometer will be used to measure vibration sense. Participants will be placed in a relaxed position in a chair and tested with the same script and application of the vibration unit to the proximal lower extremity where sensation is intact. Mid-plantar pad and the tip of the great toe will be tested via 2 trials per protocol and averaged. The amplitude is directly proportional to the square of the applied voltage and higher numbers indicate less perception of sensation.
Salivary Cortisol | Change from baseline salivary cortisol at 8 weeks
  Salivary cortisol will be collected using the Salivette device and standardized methodology with minimum invasiveness. Higher numbers indicate greater cortisol levels and higher stress

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Galantino, PT, PhD, Principal Investigator — Stockton University - Program in Physical Therapy
Locations (2):
- United States (2):
  - Leadership Studio, Atlantic City, New Jersey
  - Bacharach Institute for Rehabilitation, Pomona, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided
Will share deidentified data along with analysis to build from pilot data findings to engage in larger randomized clinical trials.

REFERENCES:
- [Background] Stout NL, Silver JK, Raj VS, Rowland J, Gerber L, Cheville A, Ness KK, Radomski M, Nitkin R, Stubblefield MD, Morris GS, Acevedo A, Brandon Z, Braveman B, Cunningham S, Gilchrist L, Jones L, Padgett L, Wolf T, Winters-Stone K, Campbell G, Hendricks J, Perkin K, Chan L. Toward a National Initiative in Cancer Rehabilitation: Recommendations From a Subject Matter Expert Group. Arch Phys Med Rehabil. 2016 Nov;97(11):2006-2015. doi: 10.1016/j.apmr.2016.05.002. Epub 2016 May 27. PMID 27237580
- [Background] Agarwal RP, Maroko-Afek A. Yoga into Cancer Care: A Review of the Evidence-based Research. Int J Yoga. 2018 Jan-Apr;11(1):3-29. doi: 10.4103/ijoy.IJOY_42_17. PMID 29343927
- [Background] Galantino ML, Greene L, Daniels L, Dooley B, Muscatello L, O'Donnell L. Longitudinal impact of yoga on chemotherapy-related cognitive impairment and quality of life in women with early stage breast cancer: a case series. Explore (NY). 2012 Mar-Apr;8(2):127-35. doi: 10.1016/j.explore.2011.12.001. PMID 22385567
- [Background] Galantino ML, Desai K, Greene L, Demichele A, Stricker CT, Mao JJ. Impact of yoga on functional outcomes in breast cancer survivors with aromatase inhibitor-associated arthralgias. Integr Cancer Ther. 2012 Dec;11(4):313-20. doi: 10.1177/1534735411413270. Epub 2011 Jul 6. PMID 21733988
- [Derived] Galantino ML, Tiger R, Brooks J, Jang S, Wilson K. Impact of Somatic Yoga and Meditation on Fall Risk, Function, and Quality of Life for Chemotherapy-Induced Peripheral Neuropathy Syndrome in Cancer Survivors. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419850627. doi: 10.1177/1534735419850627. PMID 31131640